CLINICAL TRIAL: NCT02186483
Title: An Open-label, Randomized, Multiple-dose, Crossover Study to Evaluate the Drug-drug Interaction Following Coadministration of Metformin and Rosuvastatin in Healthy Male Volunteers
Brief Title: Clinical Trial to Investigate the Pharmacokinetics Drug Interaction Between Metformin and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP_1310-P1-DI
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2014-07

CONDITIONS: Hyperlipidemia; Diabetes
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus | interventions — Metformin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin (Experimental): Metformin and Rosuvastatin: Volunteers will be taken Metformin-Rosuvastatin-Co-administration
  Interventions: Drug: Metformin; Drug: Rosuvastatin; Drug: Metformin and Rosuvastatin
- Rosuvastatin (Experimental): Metformin and Rosuvastatin: Volunteers will be taken Rosuvastatin-Co-administration-Metformin
  Interventions: Drug: Metformin; Drug: Rosuvastatin; Drug: Metformin and Rosuvastatin
- Co-administration (Experimental): Metformin and Rosuvastatin: Volunteers will be taken Co-administration-Metformin-Rosuvastatin
  Interventions: Drug: Metformin; Drug: Rosuvastatin; Drug: Metformin and Rosuvastatin

INTERVENTIONS:
Drug: Metformin — Metformin,1000mg, once daily
  Other Names: Glucodown OR SR tablet
Drug: Rosuvastatin — Rosuvastatin, 20 mg, once daily
  Other Names: Crestor tablet
Drug: Metformin and Rosuvastatin — Metformin, 1000mg, once daily Rosuvastatin, 20mg, once daily
  Other Names: Glucodown OR SR tablet and Crestor tablet

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic drug interaction between Metformin and Rosuvastatin in healthy male volunteers.

DETAILED DESCRIPTION:
Drug-drug Interaction Following Co-administration of Metformin and Rosuvastatin in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* 19~55 years healthy male
* BMI measurement 19.0kg/m^2~ 28.0kg/m^2
* Signed informed consent form from to participate voluntarily and to comply with the trial requirements.

Exclusion Criteria:

* History of clinically significant kidney, liver, gastro-intestinal system, cardiovascular system, respiratory system, tumor or blood disorders, nervous system, immune system, endocrine disorders, cardiovascular diseases, mental disorders (mood disorders, obsessive-compulsive disorder, etc.)
* SBP>140mmHg or <90mmHg, DBP>90mmHg or <60mmHg.
* An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
* History of drug abuse
* A alcohol consumer(alcohol>140g/week) or smoker(cigarette>10 cigarettes/day) Hypersensitivity reaction in history of investigational drugs or specific drugs(aspirin, antibiotics)
* Administrated investigational product in a previous clinical trial within 60 days of the screening day in this study.
* Administrated drugs which can inhibit or induce OCT2, OATP1B1 transporter within 30 days of the screening day in this study.(ex: proton pump inhibitor, rifampicin)
* Glomerular filtration rate<60mL/min
* Donated blood within 60 days prior to the screening day or apheresis blood within 30 days prior to the screening day .

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cmax,ss, AUCτ | 32h

SECONDARY OUTCOMES:
Tmax,ss | 32h
t1/2 | 32h
Cmin,ss | 32h
CL/Fss | 32h
Vd/Fss | 32h

CONTACTS AND LOCATIONS:
Overall Officials: Jung-ryul Kim, MD, Ph.D, Principal Investigator — Samsung Medical Center(SMC)
Locations (1):
- Samsung Medical Center(SMC), Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No